CLINICAL TRIAL: NCT02306473
Title: A Novel Non-invasive Way to Measure Airway Epithelial Permeability in Human Subjects
Brief Title: The Leaky Lung Test
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Syntara (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steve Nicholas Georas, Professor of Medicine, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RSRB00043414; R01HL122424 (NIH)
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Asthma; Allergy; Reactive Airway Disease; Lung Diseases, Obstructive
MeSH Terms: conditions — Asthma; Hypersensitivity; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asthma (Experimental): Subjects with asthma will be exposed to inhaled mannitol according to FDA approved protocols.
  Interventions: Drug: Mannitol
- Controls (Experimental): Healthy control subjects will be exposed to inhaled mannitol according to FDA approved protocols.
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Mannitol — Subjects will be challenged with inhaled mannitol according to already approved protocols.
  Other Names: Aridol for bronchoprovocation

SUMMARY:
This is a clinical trial designed to test the hypothesis that measuring the absorption and excretion of inhaled mannitol will provide a clinically useful marker of airway epithelial permeability in asthma.

DETAILED DESCRIPTION:
A cohort of subjects with asthma and healthy controls will be exposed to inhaled mannitol according to FDA approved protocols for bronchoprovocation. Mannitol will be measured in the bloodstream and urine and used to determine an airway permeability index. This is a proof of concept study and not a trial of new therapeutics.

ELIGIBILITY:
Inclusion criteria: Asthma The diagnosis of asthma will be based on a consistent history, physical exam, and previous physician diagnosis of asthma. Consistent historical features of asthma include episodic wheezing, shortness of breath, chest tightness, or cough, often precipitated by known environmental triggers (e.g. respiratory viral infection, exposure to pollen, exercise, or stress). Consistent physical findings of asthma include audible expiratory wheezing and findings of associated diseases (e.g. eczema, allergic rhinitis), although the physical exam may be normal in between asthma attacks. Subjects will need to be free of asthma symptoms at time of challenge testing. Most asthmatic subjects should demonstrate bronchial reactivity during the mannitol challenge test.

Inclusion criteria: Non-asthmatic controls Healthy control subjects will be recruited in order to define baseline values for serum and urine mannitol. Healthy control subjects will be defined by the lack of symptoms or physical findings of asthma or other allergic diseases (e.g. eczema, allergic rhinitis), and absence of any other chronic lung disease. Healthy subjects should also not demonstrate bronchial reactivity during a mannitol challenge test.

Exclusion Criteria:

1. >5 pack year history of tobacco use or active smoking.
2. Other chronic or active lung diseases (e.g. COPD, pulmonary fibrosis, lung cancer)
3. History of significant renal insufficiency of liver disease
4. Asthma subjects with severe disease according to NAEPP guidelines (e.g. severe ongoing symptoms despite high-dose inhaled or oral glucocorticoids)
5. Asthma subjects with a baseline FEV1<65% predicted
6. Asthma subjects unwilling or unable to withhold medications prior to testing
7. Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Airway permeability index (Urinary clearance of mannitol overtime) | 24 hours
  Urinary clearance of mannitol overtime

SECONDARY OUTCOMES:
Absorption of mannitol (Absorption and clearance of mannitol from the bloodstream) | 6 hours
  Absorption and clearance of mannitol from the bloodstream

CONTACTS AND LOCATIONS:
Overall Officials: Steve N Georas, M.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States